CLINICAL TRIAL: NCT04637633
Title: Topical Cyclosporine-A for Management of Epiphora in Eyes With Acquired Punctal Stenosis
Brief Title: Topical Cyclosporine-A for Management of Epiphora
Acronym: CSA-epiphora
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Farwaniya Hospital (Other Government)
Responsible Party: Principal Investigator, Mona A Nassief, lecturer of ophthalmology Mansoura University Egypt currentlty working as senior registrar in Farwaniya Hospital, Farwaniya Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Farwanyia Hospital
Record Dates: First submitted 2020-07-29; First posted 2020-11-20 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Epiphora
Keywords: cyclosporine A; Epiphora; punctal stenosis
MeSH Terms: conditions — Lacrimal Apparatus Diseases | interventions — Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cyclosporine A (Experimental): All patients were treated with topical 0.05% CsA (Restasis®, Allergan Inc, Irvine, California) on twice daily dose, in addition to the topical preservative free artificial tears Q.I. D.
  Interventions: Drug: topical 0.05% CsA (Restasis®, Allergan Inc, Irvine, California)twice daily dose,

INTERVENTIONS:
Drug: topical 0.05% CsA (Restasis®, Allergan Inc, Irvine, California)twice daily dose, — topical preservative free artificial tears Q.I. D.
  Other Names: preservative free artificial tears

SUMMARY:
to investigate the clinical outcomes and tolerances of Cyclosporine A (CsA) in treating epiphora in eyes with acquired punctum stenosis

DETAILED DESCRIPTION:
a prospective study included patients who were referred to our outpatient clinics in Farwanyia hospital, Kuwait during the period between July 2019 and January 2020, having symptomatic epiphora associated with severe acquired lower punctal stenosis. Patients were treated with topical 0.05% CsA on twice daily dose with topical preservative free artificial tears Q.I. D. Patients were followed up monthly for at least 3 months by epiphora grading, Fluorescein dye disappearance test (FDT) and evaluating the patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either sex
* had a diagnosis of epiphora that persisted more than three months both indoors and outdoors
* grade 0 punctal stenosis
* did not adequately respond to artificial tears, topical corticosteroids and topical antibiotics or in whom corticosteroids were discontinued due to their side effects.

Exclusion Criteria:

* congenital punctal obstruction
* edematous puncti
* allergic conjunctivitis
* history of dacryocystitis,
* inflammatory systemic diseases
* any previous chemotherapy treatment, and local irradiation.
* other causes of epiphora, lid laxity, entropion, and ectropion
* lid malposition, canalicular or nasolacrimal sac or duct obstruction
* previous eyelid or lacrimal drainage surgery
* untreated conjunctivitis or blepharitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Epiphora grading | 3 months
  Munk grading system score from 0 to 5 the higher the worse

SECONDARY OUTCOMES:
Fluorescein dye disappearance test (FDT) | 3 months
  via installing a drop of 2% fluorescein and asses the height of the tear film in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Farwanyia Hospital, Kuwait City, Farwanyia, Kuwait

IPD SHARING:
Plan to Share IPD: No